CLINICAL TRIAL: NCT00929968
Title: A Randomized, Double-blind, Placebo and Calibrator Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Intravenous Doses of VAK694 in Subjects With Seasonal Rhinitis During Natural Exposure to Allergen
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Doses of VAK694 in Atopic Subjects With Seasonal Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CVAK694A2201
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-05

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis,; atopic patients,; seasonal allergy,; ragweed allergy
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo to VAK694 (Placebo Comparator)
  Interventions: Biological: Placebo
- VAK694 (Experimental)
  Interventions: Biological: VAK694
- Fluticasone propionate (Active Comparator)
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Biological: Placebo
  Arms: Placebo to VAK694
Biological: VAK694
  Arms: VAK694
Drug: Fluticasone
  Arms: Fluticasone propionate

SUMMARY:
This study will assess the safety and tolerability of multiple doses of VAK694 as well as change in symptoms and biomarkers in patients with seasonal allergic rhinitis

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between ages of 18 to 60 in good health
* History of atopy for at least 2 years and positive skin prick test to ragweed allergen

Exclusion criteria:

* History of asthma treated with corticosteroids
* Smokers with a smoking history of > 10 pack/years or smoking in the past year
* History of chronic obstructive pulmonary disease

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of prolonged administration of multiple intravenous doses of VAK694 as well as the preliminary efficacy of multiple intravenous doses of VAK694 in atopic subjects | 12 weeks

SECONDARY OUTCOMES:
To evaluate pharmacokinetics of multiple intravenous doses of VAK694 in atopic subjects | 12 weeks
Change in serum levels of total and antigen specific IgE and total and antigen specific IgG | 12 weeks
Immunogenicity of multiple intravenous doses of VAK694 | 12 weeks
Changes in rhinitis visual-analogue score and the use of symptom relief during both the peak and entire allergy season. | 12 weeks
Changes in biomarkers of immunomodulation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Altoona Center for Clinical Research, Duncansville, Pennsylvania, United States
- Novartis Investigative Site, Ottawa, Ontario, Canada

REFERENCES:
- See also: Results for CVAK694A2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6443